CLINICAL TRIAL: NCT02258087
Title: Comparison of High-dose- Versus Low-dose-rate Brachytherapy as Monotherapy in the Treatment of Early, Organ Confined Prostate Cancer.
Brief Title: HDR vs LDR Brachytherapy as Monotherapy in the Treatment of Localized Prostate Cancer.
Acronym: PROMOBRA
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Institute of Oncology, Hungary (Other)
Responsible Party: Principal Investigator, Peter Agoston, MD, PhD, National Institute of Oncology, Hungary
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PROMOBRA-2013
Record Dates: First submitted 2014-09-30; First posted 2014-10-07 (Estimated); Last update posted 2014-10-07 (Estimated); Status verified 2014-10

CONDITIONS: Adenocarcinoma of Prostate
Keywords: Prostate, Cancer, Brachytherapy, HDR, LDR, monotherapy
MeSH Terms: conditions — Neoplasms; Barakat syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- LDRPBT (Active Comparator): Patients with low and selected intermediate risk prostate cancer are treated with Prostate LDR brachytherapy as monotherapy. 145 Gy is prescribed to the prostate. I-125 radioactive sources are used. Transperineal approach, rectal ultrasound guidance, inverse treatment planning, real time dose optimization is applied.
  Interventions: Radiation: LDR Brachytherapy
- HDRPBT (Experimental): Patients with low and selected intermediate risk prostate cancer are treated with prostate HDR brachytherapy as monotherapy. The prescribed dose is 1x19 Gy to the whole prostate. Ir-192 radioactive source is used. Transperineal approach, rectal ultrasound guidance, inverse treatment planning, real time dose optimization is applied.
  Interventions: Radiation: HDR Brachytherapy

INTERVENTIONS:
Radiation: LDR Brachytherapy — In spinal anaesthesia patients' prostate are treated with low-dose-rate or brachytherapy using transrectal ultrasound guidance. Radiation sources (iodine-125 isotopes) are implanted into the prostate through transperineal needle insertion. Real time dose planning is applied. The prescribed dose to the whole prostate is 145 Gy.
  Other Names: Seed brachytherapy; Permanent implantation prostate brachytherapy
  Arms: LDRPBT
Radiation: HDR Brachytherapy — In spinal anaesthesia patients' prostate are treated with one fraction of HDR brachytherapy. The prescribed dose to the whole prostate is 1x19 Gy. Ir-192 radioactive stepping source is used for the treatment with after-loading technique. Transperineal approach, rectal ultrasound guidance, inverse treatment planning, real time intraoperative needle position update and dose optimization is applied.
  Other Names: temporary implant
  Arms: HDRPBT

SUMMARY:
Investigators compare in a randomized clinical trial the results and side effects of high-dose- and low-dose-rate brachytherapy as monotherapy in the treatment of early, organ confined prostate cancer patients.

DETAILED DESCRIPTION:
Permanent implant prostate brachytherapy (LDRPBT) is a well established and proved method in the treatment of patients with low or selected intermediate risk, organ confined prostate cancer.

There are number of studies with high-dose rate brachytherapy (HDRPBT) as monotherapy with several fractionation schedule treating the same group of patients. One phase II trial showed its effectiveness given in one fraction of 19 Gy.

In the trial investigators randomly select patients to treat with either LDR prostate brachytherapy (145Gy) or HDR prostate brachytherapy (1x19Gy) as monotherapy.

Patients are stratified into two pretreatment group: 1. low risk, 2. selected intermediate risk group.

Brachytherapy is given in spinal anaesthesia, using transrectal ultrasound based real time treatment planning. Dose constraints are defined for both methods.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) status <=1
* 40-75 years old
* expected life expectancy>10 years
* low risk prostate cancer (Prostate specific antigen (PSA)<=10ng/ml, gleason score <7, T status<=2a), less than 50 % positive biopsy cores
* selected intermediate prostate cancer (PSA)=10-<15ng/ml or gleason score =3+4(but not 4+3), or T2b-c, less than 50 % positive biopsy cores)
* International prostate symptom score (IPSS) <=15
* Prostate volume<=50cm3
* no pubic interference
* no prior prostate operation, except biopsy
* no prior radiation to pelvis
* patient signed the informed consent

Exclusion Criteria:

* <40 years or >75 years old
* PSA>15 ng/ml gleason score 4+3 , score 8-10
* ECOG>=2
* T3-4
* percent core positivity >50 %
* TUR operation within six months prior to the brachytherapy prostate volume<10 cm3 or >50 cm3 IPSS >15

Ages: 40 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2014-09; Primary Completion 2017-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Acute side effects | 6 months
  Acute gastrointestinal, urogenital and other side effects occuring within six months after the procedure, according to the Common Toxicity Criteria for Adverse Effects (CTCAE 4.0v) scale
Chronic side effects | from 6 months to five year
  Chronic gastrointestinal, urogenital and other side effects occuring within six months after the procedure, according to the CTCAE 4.0v scale

SECONDARY OUTCOMES:
quality of life | 5 years
  Assessing patients' quality of life according to the a 25 question prostate module (PR-25) of the European Organization for Research and Treatment of Cancer quality of life questionnaire (EORTC QlQ-30).
quality of life | 5 years
  Assessing patients' quality of life according to the International Index for Erectile Function (IIEF) questionnaire
Biochemical relapse free survival (bRFS) | 5 years
  Censoring an event when biochemical relapse occurs using the American Society of Therapeutic Radiation and Oncology (ASTRO) Phoenix definition for PSA relapse (nadir + 2 ng/ml increase)
Locoregional tumor free survival | 5 years
  Censoring an event when either local or regional relapse occurs
Disease specific survival (DSS) | 5 years
  Censoring an event when patient dies due to prostate cancer

CONTACTS AND LOCATIONS:
Overall Officials: Peter Agoston, MD, PHD, Principal Investigator — NIO, Hungary
Locations (1):
- Peter Agoston, Budapest, Hungary